CLINICAL TRIAL: NCT06193928
Title: Long-Term SafEty and Clinical Outcomes of LivmArli in Patients in the United States (LEAP-US)
Acronym: LEAP
Status: Recruiting | Type: Observational
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MRX-310
Record Dates: First submitted 2023-12-11; First posted 2024-01-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Alagille Syndrome; Progressive Familial Intrahepatic Cholestasis
Keywords: ALGS; Liver Diseases; PFIC; Livmarli; Alagille Syndrome; Progressive Familial Intrahepatic Cholestasis
MeSH Terms: conditions — Alagille Syndrome; Cholestasis, progressive familial intrahepatic 1; Liver Diseases | interventions — maralixibat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Alagille syndrome (ALGS): * A clinically and/or genetically confirmed ALGS diagnosis
  * Participant prescribed Livmarli
  Interventions: Drug: Livmarli
- Progressive familial intrahepatic cholestasis (PFIC): * A clinically and/or genetically confirmed PFIC diagnosis
  * Prescribed Livmarli
  Interventions: Drug: Livmarli

INTERVENTIONS:
Drug: Livmarli — The recommended dosage is 380 mcg/kg once daily.
  Other Names: Maralixibat
  Groups: Alagille syndrome (ALGS)
Drug: Livmarli — The recommended dosage us 570 mcg/kg twice daily.
  Other Names: Maralixibat
  Groups: Progressive familial intrahepatic cholestasis (PFIC)

SUMMARY:
The objective of this 5-year, prospective, observational cohort study is to evaluate the long-term safety and clinical outcomes of patients with Alagille syndrome (ALGS) or Progressive familial intrahepatic cholestasis (PFIC) treated with Livmarli.

DETAILED DESCRIPTION:
Livmarli® is a novel, minimally absorbed, pharmacological product that inhibits the ileal bile acid transporter (IBAT) in the terminal ileum, leading to reduced levels of bile acids. Livmarli (maralixibat) has been developed by Mirum Pharmaceuticals and was the first treatment approved by the US Food and Drug Administration (FDA) for the treatment of cholestatic pruritus in patients 3 months of age and older with Alagille syndrome (ALGS). Subsequently, Livmarli was approved by the FDA for the treatment of cholestatic pruritus in patients 12 months of age and older with Progressive familial intrahepatic cholestasis (PFIC). To be eligible for the study, participants must meet the following criteria:

* A clinically and/or genetically confirmed ALGS diagnosis or PFIC diagnosis
* Prescribed Livmarli

ELIGIBILITY:
Inclusion Criteria:

* A clinically and/or genetically confirmed ALGS diagnosis or PFIC diagnosis
* Participant prescribed Livmarli

Exclusion Criteria:

* Refusal to provide informed consent/assent (if required by the local IRB)
* Previously or currently on Livmarli through participation in a clinical study or expanded access program
* Participants who have previously received an SBD or LT
* Any condition or abnormalities that, in the opinion of the investigator, may interfere with the participant participating in or completing the study
* Participants who have received an investigational drug within 30 days of the first dose of Livmarli

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with ALGS and PFIC prescribed Livmarli at a participating study center and who consent/assent to participation (if required by the local IRB/IEC) will be included in the study at the discretion of the center investigator.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2028-09-20 (Estimated); Study Completion 2030-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Long-Term Clinical Outcomes | Long-term clinical outcomes (SBD, LT, portal hypertension, all-cause mortality) up to 180 days after discontinuation of Livmarli will be recorded.
  The dates, and reasons for the following first events (of this first endpoint) will be collected: Surgical Biliary Diversion (SBD), Liver Transplant (LT), and all-cause mortality. In addition, manifestations of clinically evident portal hypertension (CEPH) will be captured during each interval event assessments.
Liver Transplant Indication and Waitlist Status | LT waitlist status will be collected at enrollment and every 6 months for 5 years.
  LT waitlist status will be collected, including when placed on or removed from LT waitlist.
Assessment of Growth and Development | Weight (kilograms) and height (centimeters) z-scores will be collected every year for 5 years.
  Height and weight will be collected both at the time the participant started Livmarli and at the time of enrollment in the study. Subsequent weight will be collected for up to 5 years.
  Weight z-score (kilograms) and height z-score (centimeters) will be assessed and reported every year for 5 years.
Incidence of Clinical Events Potentially Related to Fat-Soluble Vitamin Deficiencies and Their Long-Term Sequelae | The incidence of events will be assessed and reported every year for 5 years.
  Bleeding events (including all gastrointestinal [GI] or non-GI bleeding requiring hospitalization, emergency department care, or transfusion) and fracture events will be reported.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Children's Hospital Los Angeles CHLA, Los Angeles, California
  - Section of Gastroenterology, Hepatology and Nutrition, Department of Pediatrics and the Digestive Health Institute, Children's Hospital of Colorado and University of Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta - Emory University School of Medicine, Atlanta, Georgia
  - Children's Mercy Kansas City, Department of Gastroenterology, Section of Hepatology, Kansas City, Missouri
  - Oregon Health and Science University, Division of Pediatric Gastroenterology, Department of Pediatrics, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Division of Pediatric Gastroenterology, Hepatology and Nutrition, Salt Lake City, Utah

REFERENCES:
- See also: Mirum Pharmaceuticals homepage — https://mirumpharma.com/
- See also: Genetics Home Reference - ALGS — https://ghr.nlm.nih.gov/condition/alagille-syndrome
- See also: US FDA Resources — https://clinicaltrials.gov/ct2/info/fdalinks